CLINICAL TRIAL: NCT03967925
Title: A Randomised, Double Blind, Controlled Mechanistic Study of Rituximab and Belimumab Combination Therapy in PR3 ANCA-associated Vasculitis
Brief Title: Rituximab and Belimumab Combination Therapy in PR3 Vasculitis
Acronym: COMBIVAS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rachel Jones (Other)
Collaborators: GlaxoSmithKline (Industry); Medical Research Council (Other Government); Imperial College London (Other); University College, London (Other); Newcastle University (Other); University of Glasgow (Other); University of Cambridge (Other)
Responsible Party: Sponsor-Investigator, Rachel Jones, Consultant Nephrologist, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 206852
Record Dates: First submitted 2019-01-18; First posted 2019-05-30 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: ANCA Associated Vasculitis; Granulomatosis With Polyangiitis
Keywords: proteinase 3
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Granulomatosis with Polyangiitis | interventions — belimumab; Rituximab; Prednisolone; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Belimumab (Active Comparator): Weekly 200mg SC injections of belimumab for 12 months
  Interventions: Drug: Belimumab; Drug: Rituximab; Drug: Prednisolone
- Belimumab placebo (Placebo Comparator): Weekly SC injections of belimumab placebo for 12 months
  Interventions: Drug: Rituximab; Drug: Prednisolone

INTERVENTIONS:
Drug: Belimumab — Sub-cutaneous injection
  Other Names: Benlysta
  Arms: Belimumab
Drug: Rituximab — IV infusion 1g x 2
  Other Names: Truxima
Drug: Prednisolone — 20mg prednisolone tapering dose
  Other Names: prednisone

SUMMARY:
Mechanistic study to assess whether dual B-cell immunotherapy by co-administration of rituximab and belimumab will result in improvements in biological endpoints, functional outcomes and clinical status compared to rituximab with placebo.

DETAILED DESCRIPTION:
AAV is an organ and life threatening multisystem autoimmune disease, where ANCA are strongly implicated in disease pathogenesis, causing neutrophil activation and endothelial damage. B cell depletion with rituximab, and treatment with glucocorticoids, is associated with reduction in ANCA levels and clinical remission in AAV. However, patients with proteinase 3 (PR3) ANCA subtype and/or predominantly granulomatous disease have a lower remission rate (42% vs 9% failure rate compared to other subtypes) after rituximab and glucocorticoids, with a high subsequent relapse risk of 50% by 13 months. There is a need for newer therapies to reduce the time to remission, to spare glucocorticoid use, and to promote long-lasting remission without risk of relapse. Scientific evidence suggests that dual B-cell targeted immunotherapy with both B cell depletion (i.e. rituximab as anti-CD20) and B lymphocyte stimulator (BLyS) blockade (i.e. belimumab) may be more efficacious than targeting either mechanism alone. Therefore, this mechanistic trial will assess whether dual B-cell immunotherapy by co-administration of rituximab and belimumab will result in improvements in mechanistic endpoints, functional outcomes and clinical status compared to rituximab with placebo.

The efficacy of B cell therapy depends on depletion of pathogenic B cells and the regulated reconstitution of the B cell compartment. Response to rituximab is associated with peripheral blood B cell depletion, but this is incomplete on high resolution FACS and at the disease tissue level in ANCA vasculitis patients. Early relapse is associated with a failure to become ANCA negative by 6 months, a failure of tissue B cell depletion (including PR3 specific B cells), a high proportion of memory B cells before rituximab treatment and early peripheral B cell reconstitution with a predominant memory phenotype.

Combining B cell depleting therapy (rituximab) with BLyS antagonism (belimumab) may enhance B cell targeting in AAV through several mechanisms: belimumab reduces both CD20+ and CD20- plasmablast populations in SLE patients hence combination therapy may impact a broader B cell population than targeting CD20 alone. High BLyS levels in tissue niches may also retain B cells and protect against depletion by rituximab. As observed in the BLISS studies, belimumab is associated with an early rise in peripheral blood memory B cells, possibly due to mobilisation from lymphoid tissue. Studies on tissue B cell depletion and BLyS in pre-clinical models support the concept of combining anti-CD20 and BLyS targeting and assessing tissue depletion in lymph node biopsies as well as in blood. High BLyS levels during B cell reconstitution post rituximab can promote return of autoreactive B cell resulting in more severe flares. Regulation of BLyS levels post depletion is thought to set a higher stringency for B cell reconstitution, selecting out autoreactive B cells and would directly target any BLyS driven rebound effect.

Rituximab will be dosed at Days 8 and 22, after initiation of belimumab and discontinuation of baseline immunosuppressants. Dosing at Day 8 and Day 22 is justified by: a) separation of start times for belimumab and rituximab, thereby allowing for observation of safety events which may be attributable to starting treatment with the individual agents, and b) evidence that belimumab may mobilise B cells into the periphery making them available targets for anti-CD20 treatment, therefore, starting belimumab prior to rituximab may allow more efficient peripheral B cell depletion by rituximab. Continuing belimumab therapy for 52 weeks ensures that anti-BLyS activity continues during the critical timeframe of B cell reconstitution post rituximab (median time 8.5 to 12.6 months) reducing the potential for high levels of BLyS during this time. Assessments during follow-up after completion of beliumumab / belimumab-placebo therapy allow assessment of whether immunological and clinical remission is maintained once B cell reconstitution has taken place.

A barrier to research of B cell targeted therapy has been the difficulty in obtaining sequential cells from sites where the immune dysregulation occurs or sites of inflammation. Therefore, the inclusion of both lymph node biopsies and nasal tissue biopsies in this trial will potentially permit direct characterisation of pathogenic cells at key sites, their microenvironment and, critically, the interaction of B cells with helper T cells, the primary drivers of the abnormal immune response

ELIGIBILITY:
Inclusion Criteria:

Participants must be 18 of age

* Have a diagnosis of AAV (granulomatosis with polyangiitis or microscopic polyangiitis)
* Have PR3 ANCA positivity by ELISA at screening
* Have active disease defined by one major or three minor disease activity items on BVAS/WG
* Be capable of giving signed informed consent

Exclusion Criteria:

* MPO ANCA or anti-GBM antibody positivity by ELISA at screening
* Presence of pulmonary haemorrhage with hypoxia at screening
* Estimated glomerular filtration rate (eGFR) <30 ml/min/1.73m2 at screening
* Have an acute serious or chronic infection at screening
* Have received any B cell targeted therapy within 364 days of Day 1
* Have received any steroid injection (e.g., intramuscular [IM], intraarticular, or IV) within 60 days of Day 1 (unless given during or 14 days before screening period)
* Have received >1.5mg methylprednisolone (IV) between 14 days prior to screening and Day 1 (including Day 1).
* Have received oral prednisolone >10mg/day (or equivalent) on average over the 30 days prior to screening
* Have undetectable peripheral blood B cells at screening
* Have IgG <400mg/dl at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Time to PR3 ANCA negativity | Analysed at 24 months
  ELISA analysis at different time points to determine when PR3 ANCA can no longer be detected

SECONDARY OUTCOMES:
Proportion of participants with PR3 ANCA negativity | 2 years
  Measured by ELISA at various time points
Change from baseline of certain cell subsets | 2 years
  Measured by flow cytometry at various time points
Time to clinical remission | 2 years
  Measured by BVAS/WG
Incidence of serious adverse events (SAEs) | 2 years
  Hospitalisation or serious events

CONTACTS AND LOCATIONS:
Overall Officials: Rachel B Jones, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (6):
- United Kingdom (6):
  - Addenbrooke's Hospital, Cambridge
  - Glasgow Royal Infirmary, Glasgow
  - Imperial College London, London
  - Royal Free Hospital, London
  - Royal Freemann Hospital, Newcastle
  - Nottingham University Hospitals, Nottingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McClure ME, Gopaluni S, Wason J, Henderson RB, Van Maurik A, Savage CCO, Pusey CD, Salama AD, Lyons PA, Lee J, Mynard K, Jayne DR, Jones RB; on behalf the COMBIVAS investigators. A randomised study of rituximab and belimumab sequential therapy in PR3 ANCA-associated vasculitis (COMBIVAS): design of the study protocol. Trials. 2023 Mar 11;24(1):180. doi: 10.1186/s13063-023-07218-y. PMID 36906660
- [Derived] Serling-Boyd N, Wallace ZS. Management of primary vasculitides with biologic and novel small molecule medications. Curr Opin Rheumatol. 2021 Jan;33(1):8-14. doi: 10.1097/BOR.0000000000000756. PMID 33164993